CLINICAL TRIAL: NCT01434680
Title: A Phase 2, Randomized, Comparative, Multicenter Observer-Blind Study Evaluating the Safety and Immunogenicity of the New Liquid Formulation of Novartis Meningococcal C Conjugate Vaccine and of the Novartis Lyophilized Meningococcal C Conjugate Vaccine Manufactured at Two Different Sites, in Healthy Toddlers
Brief Title: Evaluating the Comparative Safety and Immunogenicity of Three Lots of Novartis Meningococcal C Conjugate Vaccine in Healthy Toddlers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V14_57
Record Dates: First submitted 2011-09-14; First posted 2011-09-15 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-03

CONDITIONS: Meningococcal Disease; Meningococcal Meningitis
Keywords: Meningococcal disease; vaccines; toddlers; prevention; Meningitis
MeSH Terms: conditions — Meningococcal Infections; Meningitis, Meningococcal; Meningitis

STUDY DESIGN:
Who Masked: Investigator

ARMS (3):
- MenC-CRM LIQ (Liquid Formulation) (Experimental): Subjects received 1 injection of MenC-CRM vaccine,liquid formulation.
  Interventions: Biological: MenC-CRM LIQ
- MenC-CRM ROS (Rosia) (Experimental): Subjects received 1 injection of MenC-CRM vaccine, lyophilized formulation produced with drug substance manufactured at Rosia, Italy
  Interventions: Biological: MenC-CRM ROS
- MenC-CRM EMV (Emeryville) (Active Comparator): Subjects received 1 injection of MenC-CRM vaccine, lyophilized formulation produced with drug substance manufactured at Emeryville, USA
  Interventions: Biological: MenC-CRM EMV

INTERVENTIONS:
Biological: MenC-CRM LIQ — One dose of MenC-CRM vaccine, liquid formulation
  Arms: MenC-CRM LIQ (Liquid Formulation)
Biological: MenC-CRM ROS — One dose of MenC-CRM vaccine, lyophilized formulation produced with drug substance manufactured at Rosia, Italy.
  Arms: MenC-CRM ROS (Rosia)
Biological: MenC-CRM EMV — One dose of MenC-CRM vaccine, lyophilized formulation produced with drug substance manufactured at Emeryville, USA.
  Arms: MenC-CRM EMV (Emeryville)

SUMMARY:
The study was to evaluate the safety and and immune response of each of three lots of Novartis Meningococcal C Conjugate Vaccine (MenC-CRM Liquid) when administered to Healthy Toddlers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy 12 - 23 (inclusive) month-old male or female toddlers.
2. A parent/legal guardian was given written informed consent after the nature of the study has been explained.
3. Available for both the visits scheduled in the study.
4. In good health as determined by medical history, physical examination and clinical judgment of the investigator.

Exclusion Criteria:

1. History of any meningococcal vaccine administration.
2. Previous known or suspected disease caused by N. meningitidis.
3. Household contact with and/or intimate exposure to an individual with laboratory confirmed N. meningitidis infection or colonization.
4. History of severe allergic reaction after previous vaccinations, allergy to Latex, or hypersensitivity to any component of the vaccine.
5. Significant acute or chronic infection within the previous 7 days or axillary temperature ≥38.0°C within the previous 3 days.
6. Individuals who have received antibiotics within 6 days before vaccination.
7. Known or suspected autoimmune disease or impairment/alteration of the immune system resulting from (for example):

   * Receipt of any immunosuppressive therapy at any time since birth.
   * Receipt of any immunostimulants at any time since birth.
   * Receipt of any systemic corticosteroids or chronic use of inhaled high-potency corticosteroids since birth (use of topical corticosteroids administered in limited areas of the body [for example, eczema on knees or face or elbows] is allowed).
   * Immune deficiency disorder, or known HIV infection.
8. History of seizure, any progressive neurological disease or Guillain Barré Syndrome (exception: one self-limited non-medicated febrile seizure is acceptable).
9. Known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
10. Receipt of blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation in the past 12 weeks.
11. Taken any antipyretic medication in the previous 6 hours.
12. Received any other vaccines within 30 days prior to enrollment or intent to receive any other vaccine during the study (Exception: Inactivated influenza vaccine may be administered up to 15 days prior to study immunization and no less than 15 days after study immunization).
13. Toddler's parent(s) or legal guardian(s) are not able to comprehend and to follow all required study procedures for the whole period of the study.
14. Participation in any clinical trial with another investigational product 30 days prior to first study visit or intent to participate in another clinical study during this study.
15. Family members or household members of site research staff.
16. History or any illness/condition that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subjects due to participation in the study.
17. Any serious chronic or progressive disease according to judgment of the investigator (neoplasm, insulin dependent diabetes, cardiac, renal or hepatic disease).

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 992 (Actual)
Dates: Start 2011-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis
Locations (11):
- Poland (11):
  - NZOZ Bioscience Sp zoo, Ul Czerkaska, Bydgoszcz
  - Department Infection Disease ZOZ, Dept Infection Disease ZOZ, Debica
  - Centrum Medyczne Graniczna Sp zoo, Ul Graniczna 45, Katowice
  - NZOZ HIPOKRATES IIspzoo, Ul Strzelecka 2, Krakow
  - Specjalistyczny Zespol, Ul Krysiewicza, Poznan
  - NZLA Michalkowice Jarosz i Partnerzy Spolka Lekarska, NZLA Michalkowice Jarosz Partnerzy Spolka Lekarska, Siemianowice Slaskie
  - Zespol Przychodni Specjalistycznych SP ZOZ w Tarnowie, E Szczeklik Hospital, Tarnów
  - Samodzielny Zespol Publicznych Zakladow Opieki Zdrowotnej w, Ul Prusicka 5355, Trzebnica
  - Klinika Pediatrii Centrum Medycznego Ksztalcenia Podyplomowe, Ceglowska 80, Warszawa
  - Amicur_Krystyna Lechka-Florianska i Partnerzy, Ul O Bujwida, Wroclaw
  - Wojewodzki Specjalistyczny Szpital im dr Wl Bieganskiego, Ul. Kniaziewicza 1-5, Łódź Voivodeship

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at eleven sites in Poland.
Pre-assignment Details: All enrolled subjects were included in the trial. Data from the group MenC-CRM ROS_EMV was not included in the primary and secondary analyses as these subjects were initially enrolled in group MenC-CRM ROS, but wrongly vaccinated with MenC-CRM EMV.
Groups:
- MenC-CRM LIQ: Subjects received 1 injection of MenC-CRM vaccine, liquid formulation.
- MenC-CRM ROS: Subjects received 1 injection of MenC-CRM vaccine, lyophilized formulation produced with drug substance manufactured at Rosia, Italy.
- MenC-CRM EMV: Subjects received 1 injection of MenC-CRM vaccine, lyophilized formulation produced with drug substance manufactured at Emeryville, USA.
- MenC-CRM ROS_EMV: Subjects enrolled to receive MenC-CRM ROS, but were mistakenly administered 1 injection of MenC-CRM EMV
Period: Overall Study
Arm/Group | MenC-CRM LIQ | MenC-CRM ROS | MenC-CRM EMV | MenC-CRM ROS_EMV
Started | 299 | 268 | 306 | 119
Completed | 296 | 266 | 304 | 119
Not Completed | 3 | 2 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MenC-CRM LIQ | MenC-CRM ROS | MenC-CRM EMV | MenC-CRM ROS_EMV | Total
Number analyzed (Participants) | 299 | 268 | 306 | 119 | 992
Age, Continuous [Mean (Standard Deviation); unit: Months] | 16.4 (3.4) | 16.2 (3.2) | 16.7 (3.4) | 17.2 (3.3) | 16.5 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143 | 131 | 141 | 50 | 465
  Male | 156 | 137 | 165 | 69 | 527

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Human Serum Bactericidal Activity Titers Against N Meningitidis Serogroup C 28 Days After Vaccination
Description: Immunogenicity was measured by human serum bactericidal activity (hSBA) geometric mean titers (GMTs)against N meningitidis type C, at day 29 after a single vaccination when administered to toddlers to assess the equivalence of MenC-CRM LIQ to MenC-CRM EMV and MenC-CRM ROS to MenC-CRM EMV.
Time Frame: 1 month postvaccination (day 29)
Population: Analysis was done on the per protocol (PP) set, i.e. the subjects who received the vaccine correctly; provided evaluable serum samples at the relevant time points; and had no major protocol violations as defined prior to analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenC-CRM LIQ | MenC-CRM ROS | MenC-CRM EMV
Number analyzed (Participants) | 283 | 259 | 281
Titers
  Day 1 | 2.1 [2 to 2.2] | 2.16 [2.05 to 2.26] | 2.15 [2.05 to 2.25]
  Day 29 | 9.84 [8.39 to 12] | 14 [12 to 16] | 12 [10 to 14]
Statistical Analysis 1: Comparison: MenC-CRM LIQ vs MenC-CRM EMV; The study would be considered a success if the two-sided 95% confidence intervals (CIs) for the hSBA GMT ratios comparing MenC-CRM LIQ to MenC-CRM EMV at 28 days after a single vaccination were both within the equivalence interval (0.5, 2.0); Test type: Non-Inferiority or Equivalence — The equivalence margin was (0.5, 2.0). If the two-sided 95% CI for the ratio of the hSBA GMTs at 28 days following vaccination was within this equivalence interval for each of the two coprimary comparisons, MenC-CRM LIQ and MenC-CRM EMV would be declared equivalent with respect to the immune response to the vaccines; p < 0.05, ANOVA; 95% CIs for the GMTs ratios was obtained by exponentiating difference of least square means of log10 transformed titers and both the limits of 95% CIs; hSBA GMT ratios = 0.82, 95% CI 2-sided [0.67 to 1.00]
Statistical Analysis 2: Comparison: MenC-CRM ROS vs MenC-CRM EMV; The study would be considered a success if the two-sided 95% confidence intervals (CIs) for the hSBA GMT ratios comparing MenC-CRM ROS to MenC-CRM EMV at 28 days after a single vaccination were both within the equivalence interval (0.5, 2.0); Test type: Non-Inferiority or Equivalence — The equivalence margin was (0.5, 2.0). If the two-sided 95% CI for the ratio of the hSBA GMTs at 28 days following vaccination was within this equivalence interval for each of the two coprimary comparisons,MenC-CRM ROS and MenC-CRM EMV would be declared equivalent with respect to the immune response to the vaccines; p < 0.05, ANOVA; 95% CIs for the GMTs ratios was obtained by exponentiating difference of least square means of log10-transformed titers and both the limits of 95% CIs; hSBA GMT ratios = 1.14, 95% CI 2-sided [0.92 to 1.41]

2. Secondary Outcome: Geometric Mean hSBA Titers Against N Meningitidis Serogroup C 28 Days After Vaccination
Description: Immunogenicity was measured by hSBA GMTs against N meningitidis type C, approximately 28 days (at day 29) after a single vaccination when administered to toddlers to assess the equivalence of MenC-CRM LIQ to MenC-CRM ROS.
Time Frame: 1 month postvaccination (day 29)
Population: Analysis was done on the per protocol (PP) set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenC-CRM LIQ | MenC-CRM ROS
Number analyzed (Participants) | 283 | 259
Titers
  Day 1 | 2.1 [2 to 2.2] | 2.16 [2.05 to 2.26]
  Day 29 | 9.84 [8.39 to 12] | 14 [12 to 16]
Statistical Analysis 1: Comparison: MenC-CRM LIQ vs MenC-CRM ROS; The secondary objective was to be assessed only if both primary objectives were met. Because of this, no adjustment for multiplicity was required. MenC-CRM liquid would be declared equivalent to MenC-CRM ROS if the two-sided 95% CI for the ratio of the hSBA GMTs at approximately 28 days following vaccination was within the equivalence interval (0.5, 2.0); Test type: Non-Inferiority or Equivalence — The equivalence margin was (0.5, 2.0). If the two-sided 95% CI for the ratio of the hSBA GMTs at 28 days following vaccination was within this equivalence interval, the two vaccine groups would be declared equivalent with respect to the immune response to the vaccines; p < 0.05, ANOVA; [statistical method as in outcome 1, analysis 2]; hSBA GMT ratios = 0.72, 95% CI 2-sided [0.58 to 0.89]

3. Secondary Outcome: Number Of Subjects Reporting Solicited Local And Systemic Adverse Events
Description: Safety was assessed as the number of subjects who reported solicited local and systemic adverse events following a single injection with either MenC-CRM LIQ or MenC-CRM ROS or MenC-CRM EMV.
  Safety was also assessed in subjects who mistakenly received MenC-CRM EMV instead of MenC-CRM ROS.
Time Frame: From day 1 through day 7
Population: Analysis was done on the safety dataset, i.e. the subjects in the exposed population who provided postvaccination safety data.
Measure: Number; unit: Number of subjects
Arm/Group | MenC-CRM LIQ | MenC-CRM ROS | MenC-CRM EMV | MenC-CRM ROS_EMV
Number analyzed (Participants) | 299 | 267 | 304 | 119
Number of subjects
  Any Local | 124 | 115 | 148 | 58
  Injection site Tenderness | 88 | 64 | 101 | 41
  Injection site Erythema | 222 | 200 | 211 | 81
  Injection site Induration | 252 | 227 | 236 | 88
  Any Systemic | 163 | 140 | 155 | 60
  Change in Eating habits | 87 | 68 | 83 | 26
  Sleepiness | 66 | 55 | 56 | 24
  Persistent Crying | 45 | 41 | 36 | 15
  Vomiting | 9 | 11 | 7 | 4
  Diarrhea | 42 | 30 | 34 | 17
  Irritability | 101 | 76 | 87 | 32
  Fever (≥38°C) | 20 | 11 | 18 | 13

ADVERSE EVENTS:
Time Frame: Solicited local and systemic adverse events from day 1 to 7. Serious adverse events (SAEs) and Unsolicited AEs (other than SAEs) from day 1 to day 29 (1 month after first vaccination).
Description: All Solicited AEs are classified as systematic assessment and all unsolicited AEs are classified as non-systematic assessment.
Arm/Group | MenC-CRM LIQ | MenC-CRM ROS | MenC-CRM EMV | MenC-CRM ROS_EMV
Serious Adverse Events (participants affected / at risk) | 0/299 | 3/267 | 2/304 | 1/119
Other Adverse Events (participants affected / at risk) | 252/299 | 227/267 | 236/304 | 88/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MenC-CRM LIQ (N=299) | MenC-CRM ROS (N=267) | MenC-CRM EMV (N=304) | MenC-CRM ROS_EMV (N=119)
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastroenteritis Rotavirus (Infections and infestations) | 0 | 2 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MenC-CRM LIQ (N=299) | MenC-CRM ROS (N=267) | MenC-CRM EMV (N=304) | MenC-CRM ROS_EMV (N=119)
Diarrhea (Gastrointestinal disorders) | 44 | 32 | 36 | 17
Crying (General disorders) | 45 | 41 | 36 | 15
Injection Site Erythema (General disorders) | 222 | 200 | 211 | 81
Injection Site Induration (General disorders) | 252 | 227 | 236 | 88
Injection Site Pain (General disorders) | 88 | 64 | 101 | 41
Irritability (General disorders) | 101 | 76 | 87 | 32
Somnolence (Nervous system disorders) | 66 | 55 | 56 | 24
Eating Disorder (Psychiatric disorders) | 88 | 68 | 83 | 26
Pyrexia (General disorders) | 27 | 15 | 23 | 17
Respiratory Tract Infection (Infections and infestations) | 10 | 7 | 12 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.